CLINICAL TRIAL: NCT02615028
Title: Kaohsiung Medical University Chung-Ho Memorial Hospital Institutional Review Board
Brief Title: Development of Novel Designed Force Plate for Measuring the Balance Ability for the Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: KMUH-IRB-20120807
Record Dates: First submitted 2015-11-17; First posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Force plate, Balance ability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Closed eyes double-leg stance (Other): Body relaxed with both arms naturally placed beside thighs, eyes closed for 40 seconds.
  Interventions: Other: Closed eyes double-leg stance

INTERVENTIONS:
Other: Closed eyes double-leg stance — Closed eyes double-leg stance: Body relaxed with both arms naturally placed beside thighs, eyes closed for 40 seconds.

SUMMARY:
To develop a force plate with a proper computing algorithm that can be used in the average household as well as within community care centers. An affordable price range will also be necessary.

DETAILED DESCRIPTION:
Many studies using force plates to examine the elders' balance ability for fall prevention. However, few studies compare the reliability differences among age in postural sway measurements even though many studies find significantly greater postural sway in the elder population than compared to the younger cohort. Investigation of this age difference is important for choosing variables to represent their postural sway improvement in order to determine the intervention outcome.

ELIGIBILITY:
Inclusion Criteria:

* Young adults between 20 and 25 yrs
* Seniors between 67 to 75 yrs.

Exclusion Criteria:

* Lower limb neuromuscular diseases
* Musculoskeletal injuries
* Any negative response

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Center of Pressure (COP) | 40 seconds.
  Balance means the coordination module of transferring the center of pressure (COP).

CONTACTS AND LOCATIONS:
Overall Officials: Lan Y Guo, Ph.D, Study Chair — Department of Sports Medicine, College of Medicine, Kaohsiung Medical University

REFERENCES:
- [Background] Corriveau, H, Hébert R, Prince F, Raîche M. Postural control in the elderly: an analysis of test-retest and interrater reliability of the COP-COM variable. Arch Phys Med Rehabil 82(1): 80-85, 2001 Lafond D, Corriveau H, Prince F. Postural control mechanisms during quiet standing in patients with diabetic sensory neuropathy. Diabetes Care 27(1):173-178, 2004 Tinetti ME. Factors associated with serious injury during falls by ambulatory nursing home residents. J Am Geriatr Soc 35(7): 644-648, 1987. Woollacott MH, Shumway-Cook A, Nashner LM. Aging and posture control: changes in sensory organization and muscular coordination. Int J Aging Hum Dev 23(2): 97-114, 1986. 5. Sheldon JH. The effect of age on the control of sway. Gerontol Clin (Basel). 1963; 5: 129-138.